CLINICAL TRIAL: NCT01922427
Title: Study of RNS60 on Post-operative Pain and Function in Patients Undergoing Knee Anterior Cruciate Reconstruction Surgery
Brief Title: Study of RNS60 on Pain and Function After Knee Anterior Cruciate Ligament Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07.1.1.H1
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — RNS60

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: RNS60

SUMMARY:
The purpose of this study is to see if use of RNS60 during ACL reconstruction surgery decreases pain and improves functional capacity post-operation.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Post-operative pain | 1 week
  Comparison of scores from validated pain scales from post-surgery to one week